CLINICAL TRIAL: NCT06098729
Title: Informatics-Based Digital Intervention to Promote Safe Exercise in Middle-Aged Adults With Type 1 Diabetes and Other Absolute Insulin Deficiency Diabetes - A Feasibility Study
Brief Title: Digital Exercise for Middle-Aged Adults With Type 1 Diabetes and Other Absolute Insulin Deficiency Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Exerscrip LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000035846; K01DK129441 (NIH)
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes; Latent Autoimmune Diabetes in Adults; Pancreatitis
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Latent Autoimmune Diabetes in Adults; Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Exercise (Experimental)
  Interventions: Behavioral: Digital Exercise

INTERVENTIONS:
Behavioral: Digital Exercise — A mobile application that delivers personalized encouragement and data-driven health insights based upon patterns in blood sugar, exercise, mood, and sleep, to assist people with type 1 diabetes in exercising more frequently and confidently

SUMMARY:
The challenges of living with type 1 diabetes often stand in the way of getting enough exercise. Continuous blood sugar monitoring has revolutionized type 1 diabetes care but remains underutilized to sustainably support exercise and related behaviors. This research will develop a mobile application that delivers personalized encouragement and data-driven health insights based upon patterns in blood sugar, exercise, mood, and sleep, to assist people with type 1 diabetes in exercising more frequently and confidently.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with type 1 diabetes (T1D) or other insulin deficiency diabetes (latent autoimmune disease of adulthood, diabetes secondary to pancreatitis)
* Low exercise levels
* Smartphone ownership
* English literacy
* Under regular care by a healthcare provider
* Home Broadband wireless Internet or cell phone network (≥25 mbps downloads, ≥3 mbps uploads)

Exclusion Criteria:

* Diabetic ketoacidosis not clearly related to pump site failure in past 6 months
* >1 episode of severe hypoglycemia (altered mental and/or physical status requiring assistance from another person for recovery) in past 6 months
* A1c ≥10.0%
* Resting blood pressure >160mmHg systolic or >100 mmHg diastolic
* Myocardial infarction or angina in past 12 months
* Uncontrolled arrhythmia (e.g., Afib with RVR, new onset Afib, ventricular tachycardia, escape rhythms)
* Congestive heart failure (stage 3 or 4)
* Exercise-induced asthma (not controlled on inhalers)
* Chronic obstructive pulmonary disease (requiring home oxygen)
* Renal failure
* Pregnancy
* Cognitive impairment
* Severe retinopathy or neuropathy.
* Other chronic disease or physical disability that would influence exercise intervention (e.g., recent spinal surgery)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garrett Ash, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Digital Exercise: Exercise intervention
Period: Overall Study
Arm/Group | Digital Exercise
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Digital Exercise: Digital exercise intervention
Arm/Group | Digital Exercise
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Usage
Description: Minutes of using application to exercise. 0 minutes/week is the lowest value, 150 minutes/week meets clinically recommended amounts.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Digital Exercise
Number analyzed (Participants) | 24
minutes/week | 168 (14)

2. Primary Outcome: Acceptability
Description: Likert-style survey of participant satisfaction. Responses are on a scale from 1 (very dissatisfied) to 5 (very satisfied)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Exercise
Number analyzed (Participants) | 24
score on a scale | 4.0 (0.9)

3. Primary Outcome: Accuracy
Description: Accuracy to predict lapses in exercise behavior ahead of time. 50% accuracy is the lowest possible value (ie, equivalent to random guessing), 80% accuracy is the goal of the study, and 100% accuracy would be the highest possible accuracy.
  This is the single outcome of a regression analysis across the entire sample. Being a single outcome, there is no measure of dispersion.
Time Frame: 4 weeks
Measure: Number; unit: percentage of lapses
Arm/Group | Digital Exercise
Number analyzed (Participants) | 24
percentage of lapses | 70

4. Secondary Outcome: Motivation States for Physical Activity
Description: Scale name: Cravings for Rest and Volitional Energy Expenditure (CRAVE) Construct: Transient state motivation for physical activity Scale ranges: 0 (not at all) to 100 (more than ever). Higher values represent a better outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Digital Exercise
Number analyzed (Participants) | 24
units on a scale | 60.1 (4.1)

5. Secondary Outcome: Moderate to Vigorous Physical Activity
Description: Minutes of moderate to vigorous physical activity registered by hip accelerometer. 0 minutes/week is the lowest value, 150 minutes/week meets clinically recommended amounts.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Digital Exercise
Number analyzed (Participants) | 24
minutes/week | 168 (14)

6. Secondary Outcome: Interview Themes
Description: Qualitatively-identified determinants and sequalae of motivation states for physical activity
Time Frame: 6 weeks
Measure: Number; unit: themes
Arm/Group | Digital Exercise
Number analyzed (Participants) | 24
themes | 4

ADVERSE EVENTS:
Time Frame: from consenting until end of follow-up, up to 9 weeks
Arm/Group | Digital Exercise
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 12/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digital Exercise (N=24)
Level 1 Hypoglycemia (Metabolism and nutrition disorders) | 3 (7)
Muscle, joint, ligament, or tendon injury (Musculoskeletal and connective tissue disorders) | 7
COVID (Infections and infestations) | 2 (2)
Skin irritation from wearable device (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This was a pilot study focused on feasibility and acceptability, so efficacy cannot be determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT06098729/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT06098729/ICF_001.pdf